CLINICAL TRIAL: NCT04405375
Title: Gemcitabine, Pegaspargase, Etoposide, and Dexamethasone (GPED) for Patients With Relapsed/Refractory or Advanced NK/T-cell Lymphoma : a Single Arm,Open-lable,Phase II Study
Brief Title: GPED Regimen for Relapsed/Refractory or Advanced ENKTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, JING-WEN WANG, Director of department of hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-6
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: extranodal NK/T-cell lymphoma; gemcitabine; etoposide; dexamethasone; pegaspargase; hemophagocytic syndrome
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphohistiocytosis, Hemophagocytic | interventions — Gemcitabine; pegaspargase; Etoposide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): gemcitabine 1.25g/㎡ d1, pegaspargase 2500IU/㎡ d1 (max dose =<3750IU) etoposide 75mg/㎡ d1-3 dexamethasone 20mg d1-4 repeated every 21 days, up to 6 cycles.
  Interventions: Drug: gemcitabin; Drug: Pegaspargase; Drug: Etoposide; Drug: Dexamethasone

INTERVENTIONS:
Drug: gemcitabin — 1.25g/㎡ d1, repeated every 21 days
Drug: Pegaspargase — 2500IU/㎡ d1, total dose=<3750IU, repeated every 21 days
Drug: Etoposide — 75mg/㎡ d1-3, repeated every 21 days
Drug: Dexamethasone — 20mg d1-4

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of gemcitabine, pegaspargase, etoposide, and dexamethasone (GPED) in the treatment of Relapsed/Refractory or advanced NK/T-cell lymphoma patients (ENKTCL).

DETAILED DESCRIPTION:
Pegaspargase is the cornor stone for the treatment of ENKTCL, and gemcitabine has been shown to be active in ENKTCL. For several patients with relapsed/refractory or advance ENKTCL, hemophagocytic sysdrome (HPS) occurs, and the prognosis is very poor. Studies have found that etoposide and dexamethasone may be effective in controlling HPS. Thus, this study aims to evaluate the role of gemcitabine, pegaspargase, etoposide, and dexamethasone (GPED) in the treatment of relapsed/refractory or advance ENKTCL, wishing to improve the prognosis for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology and immunohistochemistry confirmed diagnosis of NK/Tcell lymphoma according to WHO 2016 criteria.
* refractory or relapsed after initial remission, or stage III-IV de novo patients
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* General status ECOG score 0-3 points.
* The laboratory test within 1 week before enrollment meets the following conditions:
* Blood routine: Hb>80g/L, PLT>50×10e9/L.
* Liver function: ALT, AST, TBIL ≤2 times the upper limit of normal.
* Renal function: Cr is normal.
* Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking.
* Sign the informed consent form

Exclusion Criteria:

* Active infection requires ICU treatment. Concomitant HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are notexcluded.
* Significant organ dysfunction Pregnant and lactating women.
* Those who were known to be allergic to drugs in the study regimen.
* Patients with other tumors who require surgery or chemotherapy within 6 months.
* Other experimental drugs are being used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2020-03-21 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival (PFS) rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PFS is defined as date of enrollment to date of disease progression, relapse, death of any reason, or last follow-up, whichever comes first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | evaluated every 2 cycles of treamtent, up to one month after the end of treatment
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria
Complete response rate (CRR) | evaluated every 2 cycles of treamtent, up to one month after the end of treatment
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria
2-year overall survial (OS) rate | From date of enrollment until the date of death from any cause or last follow-up, assessed up to 24 months
  OS is defined as date of enrollment to date of death of any reason, or last follow-up, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No